CLINICAL TRIAL: NCT04036188
Title: Triamcinolone With Vitamin D Synergistic Efficacy in Psoriasis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 06715
Record Dates: First submitted 2019-05-17; First posted 2019-07-29 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Plaque Psoriasis; Vitamin D3
MeSH Terms: interventions — Triamcinolone; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subjects, investigators and blinded research staff will be masked until subjects start the open label part of the study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Triamcinolone Cream + Vitamin D3 (Experimental): This arm will continue to take Vitamin D3 at Week 16 to Week 28.
  Interventions: Drug: Triamcinolone; Dietary Supplement: Vitamin D3
- Triamcinolone Cream + Placebo (Placebo Comparator): Starting at Week 16, this arm will be given Vitamin D3 to take until Week 28.
  Interventions: Drug: Triamcinolone; Dietary Supplement: Vitamin D3; Drug: Placebo

INTERVENTIONS:
Drug: Triamcinolone — Triamcinolone 0.1% daily
Dietary Supplement: Vitamin D3 — 40,000 IU Vitamin D3 daily
Drug: Placebo — Placebo daily
  Arms: Triamcinolone Cream + Placebo

SUMMARY:
These studies are designed to assess the synergistic efficacy of topical 0.1% triamcinolone cream paired with 40,000 IU of oral vitamin D3 daily in treating mild to moderate psoriasis. The study is designed to have all subjects treated with triamcinolone cream (TAC) for 4 weeks, then will be randomized 1:1 into vitamin D3 or placebo for an additional 12 weeks. At that time, the study will become open-label and all subjects will be placed on (or continue) vitamin D3 for an additional 12 weeks. The study will take place over 28 weeks total.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Mild to severe plaque psoriasis (2% or greater Body Surface Area; Psoriasis Area and Severity Score of 2 or greater; Investigator Grade Assessment of mild-severe)

Exclusion Criteria:

* Currently taking medication that alters the normal ion balance of low-dose in blood.
* No calcium supplements 1 month prior to baseline (not including multivitamins).
* Unstable or uncontrolled illness, including but not limited to cerebro-cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic or psychiatric disease at screening.
* Abnormal laboratory values at screening, that in the opinion of the investigator, would potentially affect patient safety or data integrity.
* Not on systemic non-biologic therapy (including, but not limited to, oral psoralen plus ultraviolet A [photochemotherapy (PUVA)] light therapy; cyclosporine; corticosteroids; methotrexate; oral retinoids; apremilast; tofacitinib; mycophenolate mofetil; thioguanine; hydroxyurea; sirolimus; tacrolimus; azathioprine; leflunomide; fumaric acid derivatives; or 1, 25 dihydroxy vitamin D3 and analogues) within 28 days prior to baseline.
* No phototherapy (including either oral and topical PUVA light therapy, ultraviolet B, excimer laser, or self-treatment with tanning beds or therapeutic sunbathing) within 28 days prior to baseline.
* No topical treatment (including, but not limited to, corticosteroids [upper mid strength or lower potency topical steroids are permitted on the intertriginous areas and face], crisaborole, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, pimecrolimus, tacrolimus, emollients and other nonprescription topical products containing urea, >3% salicylic acid, alpha- or beta-hydroxyl acids, or medicated shampoos [for example those that contain >3% salicylic acid, corticosteroids, coal tar, or vitamin D3 analogues]) within 14 days prior to baseline.
* No biologic agents within 8 weeks or three half-lives, whichever is greater prior to baseline.
* History of renal impairment.
* History of renal stones.
* History of parathyroid abnormalities
* Osteoporosis
* History of severe arthritis
* Ongoing use of tanning bed or other UV device or excessive sunlight
* Unable to understand/complete informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in Psoriasis Area and Severity Score (PASI) from baseline | Week 28
  Subjects achieving a 50% improvement from baseline (PASI 50)
Improvement in Investigator Grade Assessment (IGA) from baseline | Week 28
  Subjects achieving a 1 point reduction from baseline
Improvement in Body Surface Area (BSA) from baseline | Week 28
  Subjects achieving a 50% reduction from baseline

SECONDARY OUTCOMES:
Change in Complete Metabolic Profile Values From Baseline Due to the Combination of Topical Triamcinolone Cream and Oral Vitamin D3 | Week 28
  Assess change through complete metabolic profile laboratory values
Change in Parathyroid Hormone Level Values From Baseline Due to the Combination of Topical Triamcinolone Cream and Oral Vitamin D3 | Week 28
  Assess change through parathyroid hormone level laboratory values
Change in 25-Hydroxyvitamin D Values From Baseline Due to the Combination of Topical Triamcinolone Cream and Oral Vitamin D3 | Week 28
  Assess change through 25-Hydroxyvitamin D laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/88/NCT04036188/ICF_000.pdf